CLINICAL TRIAL: NCT00432172
Title: "A Randomized Multicenter Phase II Trial to Evaluate the Effectiveness of Selective Neoadjuvant Treatment According to Immunohistochemical Subtype for HER2 Negative Breast Cancer Patients"
Brief Title: Selective Neoadjuvant Treatment According to Immunohistochemical Subtype for HER2 Negative Breast Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEICAM/2006-03
Record Dates: First submitted 2007-02-06; First posted 2007-02-07 (Estimated); Results first posted 2019-07-17 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
Keywords: Her2neu negative breast cancer.; Neoadjuvant treatment.
MeSH Terms: conditions — Breast Neoplasms | interventions — Epirubicin; Cyclophosphamide; Docetaxel; exemestane; Goserelin; Carboplatin

ARMS (4):
- Group 1 (Luminal A) Standard treatment (Active Comparator): Standard treatment: Epirubicin (E) 90 mg/ m2 intravenous (iv) in combination with Cyclophosphamide (C) 600 mg/ m2 iv every 21 days for 4 cycles, followed by docetaxel (D)100 mg/m2 iv every 21 days for 4 cycles.
  Interventions: Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Docetaxel
- Group 1 (Luminal A) Selective treatment (Experimental): Selective treatment:
  Postmenopausal patients: exemestane x 6 months Premenopausal patients: goserelin x 6 months + exemestane x 6 months
  Interventions: Drug: Exemestane; Drug: Goserelin
- Group 2 (Basal) Standard treatment (Active Comparator): Standard treatment: Epirubicin (E) 90 mg/ m2 intravenous (iv) in combination with Cyclophosphamide (C) 600 mg/ m2 iv every 21 days for 4 cycles, followed by docetaxel (D)100 mg/m2 iv every 21 days for 4 cycles.
  Interventions: Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Docetaxel
- Group 2 (Basal) Selective treatment (Experimental): Selective treatment: Epirubicin (E) 90 mg/ m2 intravenous (iv) in combination with Cyclophosphamide (C) 600 mg/ m2 iv every 21 days for 4 cycles, followed by docetaxel (D)100 mg/m2 iv and carboplatin (Cb) (area under the curve = 6 mg/mL) iv every 21 days for 4 cycles.
  Interventions: Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Docetaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Epirubicin
  Other Names: Ellence
  Arms: Group 1 (Luminal A) Standard treatment; Group 2 (Basal) Selective treatment; Group 2 (Basal) Standard treatment
Drug: Cyclophosphamide
  Other Names: Cytoxan
  Arms: Group 1 (Luminal A) Standard treatment; Group 2 (Basal) Selective treatment; Group 2 (Basal) Standard treatment
Drug: Docetaxel
  Other Names: Taxotere
  Arms: Group 1 (Luminal A) Standard treatment; Group 2 (Basal) Selective treatment; Group 2 (Basal) Standard treatment
Drug: Exemestane
  Other Names: aromasil
  Arms: Group 1 (Luminal A) Selective treatment
Drug: Goserelin
  Other Names: Zoladex
  Arms: Group 1 (Luminal A) Selective treatment
Drug: Carboplatin
  Other Names: Paraplatin
  Arms: Group 2 (Basal) Selective treatment

SUMMARY:
This is an open-label study that includes two substudies of random distribution. First,a sample of the primary tumor will be obtained and will be analyzed by an immunohistochemical technique to determine several markers.Depending on the expression of these markers, the patients will be characterize as group 1 (Luminal A phenotype) or group 2 (Basal phenotype) and a random assignment will be performed to standard or experimental treatment.

DETAILED DESCRIPTION:
Group 1 (Luminal A):

* Standard treatment: Epirubicin (E) 90 mg/ m2 intravenous (iv) in combination with Cyclophosphamide (C) 600 mg/ m2 iv every 21 days for 4 cycles, followed by docetaxel (D)100 mg/m2 iv every 21 days for 4 cycles.

EC x 4 -> D x 4

* Selective treatment: Postmenopausal patients: exemestane x 6 months; Premenopausal patients: goserelin x 6 months + exemestane x 6 months

Group 2 (Basal):

* Standard treatment: EC x 4 -> D x 4
* Selective treatment: E 90 mg/ m2 iv in combination with C 600 mg/ m2 iv every 21 days for 4 cycles, followed by D (75 mg/m2) and carboplatin (Cb) (area under the curve = 6 mg/mL) iv every 21 days for 4 cycles.

EC x 4 -> DCb x 4

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Breast cancer with histological diagnosis.
* Negative Human Epidermal Growth Factor Receptor 2 (HER2) tumours defined as immunohistochemistry (IHQ) 0,1+.
* No evidence of suspicion of metastatic disease.
* Age >= 18 years old.
* Performance status (Karnofsky index) >= 80 (ECOG 0,1).
* Adequate cardiac function by ECG in the previous 12 weeks.
* Hematology: neutrophils >= 1,5 x10^9/l; platelets >= 100 x10^9/l; hemoglobin >= 10 g/dl.
* Adequate hepatic function: total bilirubin <= 1x Upper Normal Limit (UNL); Aspartate aminotransferase (AST) (SGOT) and Alanine aminotransferase (ALT) (SGPT) <= 2.5 x UNL; alkaline phosphatase <= 2.5 x UNL.
* Adequate renal function: creatinine <= 1 x UNL; creatinine clearance >= 60 ml/min.
* Patients able to comply with study treatment and follow-up.
* Negative pregnancy test in the previous 14 days.

Exclusion Criteria:

* HER2 positive tumours (defined as IHQ 3+ or positive fluorescence in situ hybridization [FISH]).
* Prior systemic therapy for breast cancer (immunotherapy, hormonotherapy, chemotherapy).
* Prior treatment with anthracyclines or taxanes (paclitaxel, docetaxel) for any previous malignancy.
* Prior radiotherapy for breast cancer.
* Bilateral invasive breast cancer.
* Pregnant or lactating women.
* Previous grade >= 2 motor or sensorial neurotoxicity (National Cancer Institute Common Toxicity Criteria [NCICTC]).
* Other serious comorbidities: congestive heart failure or unstable angina; prior history of myocardial infarction in previous year; uncontrolled hypertension (HT); high risk arrhythmias; history of significant neurological or psychiatric disorders; uncontrolled active infection; active peptic ulcer; unstable diabetes mellitus; dyspnea at rest; or chronic therapy with oxygen.
* Previous or current history of neoplasms different from breast cancer, except for skin carcinoma, cervical in situ carcinoma, or any other tumor curatively treated and without recurrence in the last 10 years; ductal in situ carcinoma in the same breast; lobular in situ carcinoma.
* Chronic treatment with corticosteroids.
* Contraindications for administration of corticosteroids.
* Concomitant treatment with other therapy for cancer.
* Males.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2007-04-24 (Actual); Primary Completion 2010-09-01 (Actual); Study Completion 2010-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Hospital Miguel Servet
Locations (12):
- Spain (12):
  - Corporació Sanitaria Parc Taulí, Sabadell, Barcelona
  - Hospital Mutua de Terrassa, Terrassa, Barcelona
  - Onkologikoa, Donostia / San Sebastian, Gipuzkoa
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Centro Oncológico Regional de Galicia, A Coruña
  - Hospital General de Alicante, Alicante
  - Hospital del Mar, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital de la Princesa, Madrid
  - Hospital Clínico Universitario Virgen de la Victoria, Málaga
  - Hospital Clínico Universitario de Valencia, Valencia

REFERENCES:
- [Result] Alba E, Chacon JI, Lluch A, Anton A, Estevez L, Cirauqui B, Carrasco E, Calvo L, Segui MA, Ribelles N, Alvarez R, Sanchez-Munoz A, Sanchez R, Garcia-Asenjo JA, Rodriguez-Martin C, Escudero MJ, Albanell J. A randomized phase II trial of platinum salts in basal-like breast cancer patients in the neoadjuvant setting. Results from the GEICAM/2006-03, multicenter study. Breast Cancer Res Treat. 2012 Nov;136(2):487-93. doi: 10.1007/s10549-012-2100-y. Epub 2012 Oct 9. PMID 23053638
- [Result] Alba E, Calvo L, Albanell J, De la Haba JR, Arcusa Lanza A, Chacon JI, Sanchez-Rovira P, Plazaola A, Lopez Garcia-Asenjo JA, Bermejo B, Carrasco E, Lluch A; GEICAM. Chemotherapy (CT) and hormonotherapy (HT) as neoadjuvant treatment in luminal breast cancer patients: results from the GEICAM/2006-03, a multicenter, randomized, phase-II study. Ann Oncol. 2012 Dec;23(12):3069-3074. doi: 10.1093/annonc/mds132. Epub 2012 Jun 6. PMID 22674146
- [Result] Prat A, Lluch A, Albanell J, Barry WT, Fan C, Chacon JI, Parker JS, Calvo L, Plazaola A, Arcusa A, Segui-Palmer MA, Burgues O, Ribelles N, Rodriguez-Lescure A, Guerrero A, Ruiz-Borrego M, Munarriz B, Lopez JA, Adamo B, Cheang MC, Li Y, Hu Z, Gulley ML, Vidal MJ, Pitcher BN, Liu MC, Citron ML, Ellis MJ, Mardis E, Vickery T, Hudis CA, Winer EP, Carey LA, Caballero R, Carrasco E, Martin M, Perou CM, Alba E. Predicting response and survival in chemotherapy-treated triple-negative breast cancer. Br J Cancer. 2014 Oct 14;111(8):1532-41. doi: 10.1038/bjc.2014.444. Epub 2014 Aug 7. PMID 25101563
- [Result] Prat A, Lluch A, Turnbull AK, Dunbier AK, Calvo L, Albanell J, de la Haba-Rodriguez J, Arcusa A, Chacon JI, Sanchez-Rovira P, Plazaola A, Munoz M, Pare L, Parker JS, Ribelles N, Jimenez B, Bin Aiderus AA, Caballero R, Adamo B, Dowsett M, Carrasco E, Martin M, Dixon JM, Perou CM, Alba E. A PAM50-Based Chemoendocrine Score for Hormone Receptor-Positive Breast Cancer with an Intermediate Risk of Relapse. Clin Cancer Res. 2017 Jun 15;23(12):3035-3044. doi: 10.1158/1078-0432.CCR-16-2092. Epub 2016 Nov 30. PMID 27903675
- [Result] Alba E, Lluch A, Ribelles N, Anton-Torres A, Sanchez-Rovira P, Albanell J, Calvo L, Garcia-Asenjo JA, Palacios J, Chacon JI, Ruiz A, De la Haba-Rodriguez J, Segui-Palmer MA, Cirauqui B, Margeli M, Plazaola A, Barnadas A, Casas M, Caballero R, Carrasco E, Rojo F. High Proliferation Predicts Pathological Complete Response to Neoadjuvant Chemotherapy in Early Breast Cancer. Oncologist. 2016 Feb;21(2):150-5. doi: 10.1634/theoncologist.2015-0312. Epub 2016 Jan 19. PMID 26786263
- [Result] Chin SF, Santonja A, Grzelak M, Ahn S, Sammut SJ, Clifford H, Rueda OM, Pugh M, Goldgraben MA, Bardwell HA, Cho EY, Provenzano E, Rojo F, Alba E, Caldas C. Shallow whole genome sequencing for robust copy number profiling of formalin-fixed paraffin-embedded breast cancers. Exp Mol Pathol. 2018 Jun;104(3):161-169. doi: 10.1016/j.yexmp.2018.03.006. Epub 2018 Mar 31. PMID 29608913
- [Result] Santonja A, Sanchez-Munoz A, Lluch A, Chica-Parrado MR, Albanell J, Chacon JI, Antolin S, Jerez JM, de la Haba J, de Luque V, Fernandez-De Sousa CE, Vicioso L, Plata Y, Ramirez-Tortosa CL, Alvarez M, Llacer C, Zarcos-Pedrinaci I, Carrasco E, Caballero R, Martin M, Alba E. Triple negative breast cancer subtypes and pathologic complete response rate to neoadjuvant chemotherapy. Oncotarget. 2018 May 29;9(41):26406-26416. doi: 10.18632/oncotarget.25413. eCollection 2018 May 29. PMID 29899867
- [Result] Ocana A, Chacon JI, Calvo L, Anton A, Mansutti M, Albanell J, Martinez MT, Lahuerta A, Bisagni G, Bermejo B, Semiglazov V, Thill M, Chan A, Morales S, Herranz J, Tusquets I, Chiesa M, Caballero R, Valagussa P, Bianchini G, Alba E, Gianni L. Derived Neutrophil-to-Lymphocyte Ratio Predicts Pathological Complete Response to Neoadjuvant Chemotherapy in Breast Cancer. Front Oncol. 2022 Feb 11;11:827625. doi: 10.3389/fonc.2021.827625. eCollection 2021. PMID 35223459
- See also: Spanish Breast Cancer Research Group (GEICAM) is a Spanish Breast Cancer Research Group — http://www.geicam.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 (Luminal A) Standard Treatment; Group 2 (Basal) Standard Treatment: Epirubicin (E) 90 mg/ m2 intravenous (iv) in combination with Cyclophosphamide (C) 600 mg/ m2 iv every 21 days for 4 cycles, followed by docetaxel (D)100 mg/m2 iv every 21 days for 4 cycles.
- Group 1 (Luminal A) Selective Treatment: Postmenopausal patients: exemestane x 6 months Premenopausal patients: goserelin x 6 months + exemestane x 6 months
- Group 2 (Basal) Selective Treatment: Epirubicin (E) 90 mg/ m2 intravenous (iv) in combination with Cyclophosphamide (C) 600 mg/ m2 iv every 21 days for 4 cycles, followed by docetaxel (D)100 mg/m2 iv and carboplatin (Cb) (area under the curve = 6 mg/mL) iv every 21 days for 4 cycles.
Period: Overall Study
Arm/Group | Group 1 (Luminal A) Standard Treatment | Group 1 (Luminal A) Selective Treatment | Group 2 (Basal) Standard Treatment | Group 2 (Basal) Selective Treatment
Started | 47 | 48 | 46 | 48
Completed | 41 | 41 | 35 | 41
Not Completed | 6 | 7 | 11 | 7
Not completed — Physician Decision | 0 | 0 | 2 | 0
Not completed — Adverse Event | 4 | 2 | 4 | 3
Not completed — Disease progression | 0 | 2 | 5 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 2
Not completed — No treatment received | 2 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (Luminal A) Standard Treatment | Group 1 (Luminal A) Selective Treatment | Group 2 (Basal) Standard Treatment | Group 2 (Basal) Selective Treatment | Total
Number analyzed (Participants) | 47 | 48 | 46 | 48 | 189
Age, Continuous [Median (Full Range); unit: years] | 51 [32 to 74] | 50.5 [33 to 72] | 47 [27 to 70] | 47 [28 to 75] | 49 [27 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 48 | 46 | 48 | 189
  Male | 0 | 0 | 0 | 0 | 0
Menopausal status [Count of Participants; unit: Participants]
  Premenopausal | 24 | 27 | 33 | 29 | 113
  Postmenopausal | 23 | 21 | 13 | 19 | 76
Eastern Cooperative Oncology Group (ECOG) status [Count of Participants; unit: Participants] — Measure Description: ECOG score runs from 0 to 5, with 0 denoting perfect health and 5 death.
  0 - Asymptomatic
  1. - Symptomatic but completely ambulatory
  2. - Symptomatic, <50% in bed during the day
  3. - Symptomatic, >50% in bed, but not bedbound
  4. - Bedbound
  5. - Death
  Participants
    ECOG 0 | 43 | 47 | 38 | 44 | 172
    ECOG 1 | 4 | 1 | 7 | 4 | 16
    ECOG Unknown | 0 | 0 | 1 | 0 | 1
Histologic type [Count of Participants; unit: Participants]
  Ductal | 38 | 39 | 39 | 41 | 157
  Lobular | 4 | 5 | 0 | 0 | 9
  Other | 5 | 4 | 7 | 7 | 23
Histological grade [Count of Participants; unit: Participants] — Cancer cells are given a Grade (G) when they are removed from the breast and checked under a microscope. The G is based on how much the cancer cells look like normal cells.
  G1 or well differentiated (score 3, 4, or 5): cells are slower-growing, and look more like normal breast tissue.
  G2 or moderately differentiated (score 6, 7): cells are growing at a speed of and look like cells somewhere between G1 and 3.
  G3 or poorly differentiated (score 8, 9): cells look very different from normal and will probably grow and spread faster.
  Participants
    Grade 1 | 11 | 11 | 1 | 2 | 25
    Grade 2 | 30 | 27 | 9 | 13 | 79
    Grade 3 | 6 | 10 | 36 | 33 | 85
Tumor size [Count of Participants; unit: Participants] — Tumor (T) size describes the size of the tumour. Larger T is associated with inferior survival.
  TX: can't be assessed. Tis: ductal carcinoma in situ. T1: tumour is 2 centimetres (cm) across or less. T1mi: tumour is 0.1cm across or less T1a: tumour >0.1 cm but <0.5 cm T1b: tumour >0.5 cm but <1 cm T1c: tumour >1 cm but <2 cm T2: tumour >2 cm but <5 cm across. T3: tumour >5 cm across. T4a: tumour has spread into the chest wall T4b: tumour has spread into the skin and the breast might be swollen T4c: tumour has spread to both the skin and the chest wall T4d: inflammatory carcinoma
  Participants
    T1 | 1 | 1 | 3 | 6 | 11
    T2 | 36 | 34 | 34 | 31 | 135
    T3 | 10 | 13 | 8 | 10 | 41
    T4 | 0 | 0 | 1 | 1 | 2
Nodal status [Count of Participants; unit: Participants] — Node (N) describes whether the cancer has spread to the Lymph Nodes (LN). Prognosis is better when cancer has not spread to the LN. The more LN that contain cancer, the poorer prognosis tends to be.
  NX: LN can't be assessed N0: no Cancer Cells (CC) N1: CC in the LN in the armpit but the nodes are not stuck to surrounding tissues.
  N2a: CC in the LN in the armpit, which are stuck to each other and to other structures.
  N2b: CC in the LN behind the breast bone. N3a: CC in LN below the collarbone. N3b: CC in LN in the armpit and behind the breastbone. N3c: CC in LN above the collarbone.
  Participants
    N0 | 24 | 28 | 21 | 24 | 97
    N1 | 22 | 19 | 22 | 20 | 83
    N2 | 1 | 1 | 3 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Pathological Response for Basal Group 2
Description: This primary outcome only applies for the basal group 2 as per protocol. The pathological response in luminal group 1 was not pre-specified even as a Secondary Outcome. Pathological response was assessed after surgery, according to the Miller & Payne criteria, which stratifies the responses based on the proportion of remaining tumor and post-chemotherapy changes, evaluating separately the response in breast and axilla. Grades 1-4 are categorised as a partial pathological response (pPR) and grade 5 was a complete pathological response (cPR).
Time Frame: Up to 24 weeks
Population: For Group 2 (Basal) selective treatment: there was one patient who did not receive treatment, because of this is not included on the final analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2 (Basal) Standard Treatment | Group 2 (Basal) Selective Treatment
Number analyzed (Participants) | 46 | 47
Participants
  Grade 5 | 16 | 14
  Grade 4 | 5 | 11
  Grade 3 | 11 | 8
  Grade 2 | 8 | 9
  Grade 1 | 5 | 4
  Not available | 1 | 1

2. Secondary Outcome: Clinical Response Rate
Description: Clinical Response Rate was measured according to the Response Evaluation Criteria in Solid Tumors (RECIST) Criteria for target lesions before surgery: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Luminal A) Standard Treatment | Group 1 (Luminal A) Selective Treatment | Group 2 (Basal) Standard Treatment | Group 2 (Basal) Selective Treatment
Number analyzed (Participants) | 47 | 48 | 46 | 47
Participants | 31 | 23 | 32 | 36

3. Secondary Outcome: Breast Conservative Surgery Rate
Description: All patients will undergo surgery within the expected period from the end of treatment with neoadjuvant therapy. The chosen surgical option will be collected in the Case Report Form (CRF) before starting the neoadjuvant treatment, depending on the characteristics Clinics of the patient at that time (conservative surgery or mastectomy). This information will be compared with definitive surgery, to analyze whether neoadjuvant treatment has contributed to increase the rate of conservative surgery.
Time Frame: Up to 24 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Luminal A) Standard Treatment | Group 1 (Luminal A) Selective Treatment | Group 2 (Basal) Standard Treatment | Group 2 (Basal) Selective Treatment
Number analyzed (Participants) | 47 | 48 | 46 | 47
Participants
  Breast conservative surgery | 22 | 27 | 31 | 34
  Non Breast conservative surgery | 23 | 17 | 15 | 13
  Not available | 2 | 4 | 0 | 0

4. Secondary Outcome: Axillary Node Status at the Time of Surgery
Description: All the patients underwent lymphadenectomy in the foreseen term from the end of the treatment with neoadjuvant therapy, except for patients who underwent the technique of Sentinel lymph node with negative result before the start of the study treatment.
  Clinical lymph node involvement were collected in the CRF. Behind the lymphadenectomy, the rate of patients with affected lymph nodes, regardless of the type of response in the breast. To help find out if the cancer has spread outside the breast, one or more of the lymph nodes in the axilla (axillary lymph nodes) are removed for examination under a microscope. This is an important part of the determination of the stage. When the lymph nodes have cancer cells, there is a greater chance that the cancer cells have spread to other parts of the body. Decisions about treatment will depend on whether there is cancer in the lymph nodes.
Time Frame: Up to 24 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Luminal A) Standard Treatment | Group 1 (Luminal A) Selective Treatment | Group 2 (Basal) Standard Treatment | Group 2 (Basal) Selective Treatment
Number analyzed (Participants) | 47 | 48 | 46 | 47
Participants
  Negative nodes | 15 | 14 | 31 | 32
  No Negative nodes | 29 | 28 | 13 | 13
  Not available | 3 | 6 | 2 | 2

ADVERSE EVENTS:
Time Frame: Through study treatment up to surgery, an average of 21 weeks
Description: For Group 2 (Basal) selective treatment: there was one patient who did not receive treatment, because of this is not included on the final analysis.
  For Group 1 (Luminal A) Standard Treatment: there were two patients who did not receive treatment, because of this, are not included on the final analysis.
  For Group 1 (Luminal A) Selective Treatment: there were two patients who did not receive treatment, because of this, are not included on the final analysis.
Arm/Group | Group 1 (Luminal A) Standard Treatment | Group 1 (Luminal A) Selective Treatment | Group 2 (Basal) Standard Treatment | Group 2 (Basal) Selective Treatment
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/46 | 0/46 | 0/47
Serious Adverse Events (participants affected / at risk) | 5/45 | 0/46 | 16/46 | 9/47
Other Adverse Events (participants affected / at risk) | 45/45 | 46/46 | 46/46 | 47/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (Luminal A) Standard Treatment (N=45) | Group 1 (Luminal A) Selective Treatment (N=46) | Group 2 (Basal) Standard Treatment (N=46) | Group 2 (Basal) Selective Treatment (N=47)
Febrile neutropenia (Infections and infestations) | 3 | 0 | 5 | 4 — Grade 3
Pancreatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 — Acute
Infection pulmonary/ Upper airway NOS (Infections and infestations) | 1 | 0 | 0 | 0 — Grade 2
Febrile neutropenia (Infections and infestations) | 0 | 0 | 1 | 0 — Grade 4
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 0 | 0 | 2 | 3 — Grade 4
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 — Grade 3
Infection - Port a cath infection (Infections and infestations) | 0 | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 — Grade 3
Infection - Lung (pneumonia) (Infections and infestations) | 0 | 0 | 1 | 0 — Grade 3
Infection - septic shock (Infections and infestations) | 0 | 0 | 1 | 0
Mucositis/stomatitis and Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 — Mucositis grade 2, Vomiting grade 3
Diabetes decompensation (Endocrine disorders) | 0 | 0 | 1 | 0
Growth and abcessification of the tumor and cellulitis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Infection with unknown ANC - Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Surgical intervention at left upper extremity (Investigations) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (Luminal A) Standard Treatment (N=45) | Group 1 (Luminal A) Selective Treatment (N=46) | Group 2 (Basal) Standard Treatment (N=46) | Group 2 (Basal) Selective Treatment (N=47)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 5 | 0 | 2 | 4 — Grade 3
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1 | 0 | 2 | 2 — Grade 4
Lymphopenia (Blood and lymphatic system disorders) | 5 | 0 | 1 | 4 — Grade 3
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 5 | 0 | 7 | 3 — Grade 3
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 2 | 0 | 3 | 5 — Grade 4
Fatigue (General disorders) | 4 | 0 | 7 | 5 — Grade 3
Mucositis/stomatitis (Gastrointestinal disorders) | 3 | 0 | 0 | 1 — Grade 3
Febrile neutropenia (Infections and infestations) | 3 | 0 | 4 | 5 — Grade 3
ALT, SGPT (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 — Grade 3
GGT (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 — Grade 3
GGT (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 — Grade 4
Irregular menses (Reproductive system and breast disorders) | 1 | 8 | 0 | 0 — Grade 3
Febrile neutropenia (Infections and infestations) | 0 | 0 | 3 | 0 — Grade 4
Hypersensitivity (Immune system disorders) | 1 | 0 | 2 | 1 — Grade 3
Hemoglobin (Blood and lymphatic system disorders) | 0 | 0 | 0 | 4 — Grade 3
Hemoglobin (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 — Grade 4
Platelets (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 — Grade 4
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 2 — Grade 3
Vomiting (Gastrointestinal disorders) | 1 | 0 | 2 | 1 — Grade 3
Infection (Infections and infestations) | 1 | 0 | 4 | 3 — Grade 3
Hemoglobin (Blood and lymphatic system disorders) | 24 | 3 | 23 | 17 — Grade 1
Hair loss/alopecia (Skin and subcutaneous tissue disorders) | 34 | 0 | 29 | 29 — Grade 2
Hot flashes/flushes (Endocrine disorders) | 4 | 14 | 1 | 3 — Grade 1
ALT, SGPT (Metabolism and nutrition disorders) | 16 | 9 | 7 | 7 — Grade 1
Fatigue (General disorders) | 20 | 8 | 14 | 14 — Grade 1
Headache (Nervous system disorders) | 7 | 5 | 0 | 0 — Grade 1
Dizziness (General disorders) | 8 | 5 | 0 | 0 — Grade 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less